CLINICAL TRIAL: NCT01909232
Title: A Prospective, Double-Blind, Randomized, Parallel-Group, Sham-Controlled Feasibility Trial of Multi-Coil Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Major Depressive Disorder
Brief Title: A Clinical Trial for the Treatment of Depression With Repetitive Transcranial Magnetic Stimulation (rTMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cervel Neurotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN-CFS-TRMD-2
Record Dates: First submitted 2013-07-22; First posted 2013-07-26 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Depressive Disorder; Major depression; Major depressive disorder; MDD; Treatment resistant depression; Treatment intolerant depression; TRMD; TIMD; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active rTMS treatment (Experimental): Active Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator
  Interventions: Device: Active Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator
- Sham rTMS treatment (Sham Comparator): Inactive Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator
  Interventions: Device: Inactive Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator

INTERVENTIONS:
Device: Active Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator — The Cervel Neurotech multi-coil transcranial magnetic stimulator is an investigational repetitive transcranial stimulation (rTMS) device. In the active group, magnetic power output will be delivered to the subject through the coils.
  Arms: Active rTMS treatment
Device: Inactive Cervel Neurotech Multi-Coil Transcranial Magnetic Stimulator — The Cervel Neurotech multi-coil transcranial magnetic stimulator is an investigational repetitive transcranial stimulation (rTMS) device. In the inactive group, no magnetic power output will be delivered to the subject through the coils.
  Arms: Sham rTMS treatment

SUMMARY:
The purpose of this study is to determine whether the Cervel Neurotech rTMS device is safe and effective in the treatment of depression in people who do not get better with antidepressant medications or cannot take antidepressant medications.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive disorder (MDD)
* Resistance or intolerance to antidepressant medication in the current depressive episode, or intolerance to antidepressant medication in a past depressive episode
* On a stable psychotropic regimen prior to screening and be willing to maintain the current regimen and dosing for the duration of the study
* Weight less than 350 pounds

Exclusion Criteria:

* Current major depressive disorder episode of more than three years
* Seizure disorder
* History of brain injury, stroke or active central nervous system disease
* Cardiac pacemaker, implanted device (deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord unless deemed MRI-safe
* Active suicidal intent or plan
* Other significant psychiatric disorder
* Alcohol or substance dependence or abuse
* Prior treatment with transcranial magnetic stimulation
* Have failed to clinically remit to an adequate trial of electroconvulsive therapy or vagus nerve stimulation
* If female, pregnant or lactating or planning to become pregnant within the next three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in depression severity | Baseline to four weeks (the conclusion of rTMS treatment)
  Measured by the 24-item Hamilton Rating Scale for Depression

SECONDARY OUTCOMES:
Change in depression severity | Baseline to eight weeks (four weeks after the conclusion of rTMS treatment)
  Measured by the 24-item Hamilton Rating Scale for Depression
Clinically significant response | Baseline to four weeks (the conclusion of rTMS treatment)
  Defined as greater than or equal to 50% decrease in the 24-item Hamilton Rating Scale for Depression score
Clinically significant response | Baseline to eight weeks (four weeks after the conclusion of rTMS treatment)
  Defined as greater than or equal to 50% decrease in the 24-item Hamilton Rating Scale for Depression score
Remission from depression | Baseline to four weeks (the conclusion of rTMS treatment)
  Defined as 24-item Hamilton Rating Scale for Depression score less than or equal to 10
Remission from depression | Baseline to eight weeks (four weeks after the conclusion of rTMS treatment)
  Defined as 24-item Hamilton Rating Scale for Depression score less than or equal to 10
Change in quality of life | Baseline to four weeks (the conclusion of rTMS treatment)
  Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form
Change in quality of life | Baseline to eight weeks (four weeks after the conclusion of rTMS treatment)
  Measured by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form
Incidence of treatment-emergent adverse events and serious adverse events | Baseline to eight weeks (four weeks after the conclusion of rTMS treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Stannard, BS, CCRP, CCRC, Study Director — Cervel Neurotech
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - Sheppard-Pratt Health System, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Butler Hospital, Providence, Rhode Island
  - CRI Lifetree, Salt Lake City, Utah

REFERENCES:
- See also: Sponsor Website — http://www.cervel.com